CLINICAL TRIAL: NCT00308867
Title: Photodynamic Therapy With PD P 506 A or Its Placebo Compared With Cryosurgery for the Treatment of Mild to Moderate Actinic Keratosis
Brief Title: PD P 506 A-PDT Versus Placebo-PDT and Cryosurgery for the Treatment of AK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: photonamic GmbH & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK 04; EudraCT No. 2005-003556-36
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Actinic Keratosis
Keywords: PDT; AK; Cryosurgery
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Photodynamic Therapy
Procedure: Cryosurgery

SUMMARY:
The aim of this study is to investigate how the efficacy and tolerability of PD P 506 A-PDT relate to the commonly used cryosurgery in the treatment of mild to moderate AK lesions located on the head. To be able to quantify the effect the patient will be allocated to one of three treatments: PD P 506 A-PDT, cryosurgery or placebo-PDT.

DETAILED DESCRIPTION:
Actinic keratosis (AK) is a pre-cancerous skin abnormality usually caused by sun exposure. Actinic keratoses occur most commonly in fair skin, especially in the elderly. They mainly occur in sun-exposed skin areas like head and hands. It is standard of care to remove AK when diagnosed, which can be achieved by either physical ablation, chemotherapeutic agents or photodynamic therapy (PDT). In Europe, cryosurgery is the method primarily used and will therefore serve as comparator therapy for PD P 506 A-PDT. A placebo control will be necessary to validate the test system. While the comparison of PD P 506 A-PDT and cryosurgery is an open comparison, placebo-PDT and PD P 506 A-PDT will be allocated in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Caucasians
* Age > 18 years
* Diagnosis of actinic keratosis (AK) with at least four locally separated lesions located on head and/or face (hairless areas)
* Selected AK study lesions have clearly defined margins and are mild to moderate (grades I or II)
* The distance between the study lesion borders is > 1.0 cm
* Maximum diameter of each study lesion is 1.8 cm
* Skin sun sensitivity type I to IV according to Fitzpatrick

Exclusion Criteria:

* PDT Non-responder
* Pre-treatment of the AK lesions eligible for study procedures with pharmaceuticals approved for the treatment of AK during the 4 weeks preceding study treatment
* Pre-treatment of the AK lesions eligible for study procedures during the 2 weeks preceding study treatment with keratolytic agents e.g. TCA, urea or salicylic acid containing formulations
* Pre-treatment with hypericin during the 2 weeks preceding study therapy
* Treatment with systemic retinoids during the 3 months preceding study therapy
* Treatment with cytostatics or radiation during the 3 months preceding study therapy
* Female patients of childbearing potential
* Patients with clinically relevant suppression of the immune system
* Diagnosis of Porphyria
* Skin diseases that might interfere with response evaluation of study treatment
* Skin sun sensitivity type V or VI according to Fitzpatrick
* Known intolerance to one or more of the ingredients of the study medication
* Known adverse reactions to cryosurgery (including cold urticaria and cold intolerance)
* Dementia or psychic condition that might interfere with the ability to understand the study and thus give a written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding inclusion
* Suspected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Complete clinical clearance rate (CCR) of treated actinic keratosis lesions 12 weeks after study treatment. | 12 weeks

SECONDARY OUTCOMES:
CCR on patient basis 12 weeks, 6, 9 and 12 months after study treatment | 12 months
CCR of treated actinic keratosis lesions 6, 9 and 12 months after study treatment | 12 months
Adverse events/reactions and local reactions during application of the study medication as well as during and after study therapy (PDT or cryosurgery) | 12 months
Satisfaction and independent cosmetic rating of the cleared study lesions by patient and investigator in case of no recurrence of the lesion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Marcus Szeimies, Professor MD, Principal Investigator — Klinikum der Universität Regensburg, Kinik und Poliklinik für Dermatologie
Locations (26):
- Germany (26):
  - Gemeinschaftspraxis Dr. Popp, Dipl.-Med. Weber, Augsburg
  - Klinik für Dermatologie, Venerologie und Allergologie der Charite, Universitätsmedizin Berlin, Berlin
  - Praxis Dr. Simon, Berlin
  - Gemeinschaftspraxis Dres. Steinert, Biberach
  - Elbekliniken Dermatologisches Zentrum, Buxtehude
  - Gemeinschaftspraxis Dr. Dominicus, Dr. Bockhorst, Dülmen
  - Zentrum Dermatologie und Venerologie, Klinikum und Fachbereich Medizin, Frankfurt a.M.
  - Gemeinschaftspraxis Prof. Melnik, H. Hariry, Gütersloh
  - Gemeinschaftspraxis PD Dr. Petering, Dr. Röhrig-Petering, Hildesheim
  - Gemeinschaftspraxis Dr. Denzer-Fürst, Dr. Kietzmann, Kiel
  - Gemeinschaftspraxis Dr. Schirren, Dr. Lischner, Dr. Podszuweit, Kiel
  - Tagesklinik für Allergie- u. Hautkrankheiten, Kiel
  - Praxis Dr. Habermann, Koblenz
  - Praxis Dr. Fritz, Landau
  - Gemeinschaftspraxis PD Dr. Plötz, Prof. Dr. Abeck, München
  - Praxis Dr. Tanner, Nördlingen
  - Praxis Dr. Nickel, Pfungstadt
  - Praxis Dr. Itschert, Pinneberg
  - Praxis Dr. Rozsondai, Radolfzell
  - Praxis Dr. Gehse, Rastatt
  - Klinikum der Universität Regensburg, Klinik und Poliklinik für Dermatologie, Regensburg
  - Praxis Dr. Karl, Soest
  - Praxis Dr. Datz, Tübingen
  - Gemeinschaftspraxis Dr. Borrosch, Dr. Jasnoch, Vechta
  - Praxis Dr. Imberger, Westerland
  - Praxis PD Dr. Dirschka, Wuppertal